CLINICAL TRIAL: NCT01151644
Title: Safety and Efficacy of Anti-Pandemic H1N1 Vaccination in Rheumatic Diseases
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: ELOISA BONFÁ, RHEUMATOLOGY DIVISION, HOSPITAL DAS CLINICAS DA FACULDADE DE MEDICIAN DA UNIVERSIDADE DE SÃO PAULO
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEDMAC-H1N1
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-04

CONDITIONS: Rheumatoid Arthritis; Spondyloarthritis; Systemic Lupus Erythematosus (SLE); Dermatomyositis (DM); DMixed Connective Tissue Disease; Systemic Vasculitis; Systemic Sclerosis (SSc); Sjögren's Syndrome; Antiphospholipid Syndrome; Juvenile Idiopathic Arthritis; Juvenile SLE; Juvenile DM
Keywords: H1N1 VACCINE; INFLUENZA; RHEUMATIC DISEASES; ANTI-H1N1 IMMUNIZATION
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Lupus Erythematosus, Systemic; Dermatomyositis; Systemic Vasculitis; Scleroderma, Systemic; Sjogren's Syndrome; Antiphospholipid Syndrome; Arthritis, Juvenile; Influenza, Human; Rheumatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VACCINATION OF PATIENTS (Active Comparator)
  Interventions: Biological: Anti-pandemic H1N1 influenza vaccine
- VACCINATION OF HEALTHY CONTROLS (Active Comparator)
  Interventions: Biological: Anti-pandemic H1N1 influenza vaccine

INTERVENTIONS:
Biological: Anti-pandemic H1N1 influenza vaccine — inactivated, NON-adjuvanted pandemic H1N1 influenza vaccine (A/California/7/2009)

SUMMARY:
The prognosis of rheumatic diseases has improved considerably with development of therapy. However, infections are considered the most important cause of morbidity and mortality in this group of patients. One of the ways to prevent such complications is vaccination. In 2009, a new pandemic strain of influenza virus (A/H1N1/2009) has emerged raising major concerns for public health. Patients under immunosuppressive therapy have indication for immunization against influenza virus H1N1. There are, however, concerns about possibility of reactivation of autoimmune diseases, determine adverse events and insufficient immunogenicity in these patients. The lack of studies evaluating the efficacy and safety of the vaccine against influenza A(H1N1)/2009 in these rheumatic patients led to the development of this research. The objectives of this study are to evaluate the humoral response and safety of the vaccine virus A(H1N1)/2009 in immunosuppressed patients with rheumatic diseases compared to healthy controls. We have recruited 400 patients with rheumatoid arthritis, 350 with spondyloarthritis, 1000 with systemic lupus erythematosus (SLE), 150 with dermatomyositis (DM), 100 with mixed connective tissue disease, 150 with systemic vasculitis, 250 with systemic sclerosis (SSc) , 100 with Sjögren's syndrome, 100 with antiphospholipid syndrome, 100 patients with juvenile idiopathic arthritis, 80 with juvenile SLE, and 80 with juvenile DM, followed at our Rheumatology Outpatient Division and Unit Pediatric Rheumatology Children's Institute, HC-FMUSP. The control group was recruited were 200 healthy employees of ICHC-FMUSP. Informed consent was obtained from all participants and the study was approved by the Local Ethical Committee. All subjects were vaccinated against influenza virus A/(H1N1)/2009 (vaccine approved and supplied by Instituto Butantan-São Paulo). Blood samples was collected to measure levels of antibodies inhibiting hemagglutination by influenza virus A (H1N1)/2009 immediately prior to vaccination and 21 to 28 days after vaccination., Participants fulfilled a questionnaire on the immediate side effects of the vaccine. All patients with rheumatoid arthritis, spondyloarthritis, SLE, DM, systemic vasculitis, juvenile idiopathic arthritis, juvenile SLE, and DM were assessed before and 21 days after vaccination for clinical, laboratory parameters of disease activity as well as treatment. Continuous variables will be compared by t-test to evaluate differences between patients with rheumatic diseases versus healthy controls. Differences between categorical variables will be evaluated using the chi-square or Fisher exact test. Statistical significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatic diseases according to international criteria of each disorder

Exclusion Criteria:

* Previous and confirmed infection by virus A(H1N1)/2009
* History of anaphylatic reaction to egg components
* Acute fever
* Guillain-Barré syndrome, heart failure (classes III or IV), demyelinating disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-07 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse effects) and efficacy (serconversion rate) after 21 days from the vaccination | Before and after 21 days from vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology Division of Hospital das Clínicas da Faculdade de Medicina da Universidade de são PAulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Sampaio-Barros PD, Andrade DCO, Seguro LCP, Pasoto SG, Viana VST, Ribeiro ACM, Aikawa NE, Timenetsky MDCS, Precioso AR, Silva CA, Bonfa E. Pandemic non-adjuvanted influenza A H1N1 vaccine in a cohort of patients with systemic sclerosis. Rheumatology (Oxford). 2018 Oct 1;57(10):1721-1725. doi: 10.1093/rheumatology/kex330. PMID 28968874
- [Derived] de Medeiros DM, Silva CA, Bueno C, Ribeiro AC, Viana Vdos S, Carvalho JF, Bonfa E. Pandemic influenza immunization in primary antiphospholipid syndrome (PAPS): a trigger to thrombosis and autoantibody production? Lupus. 2014 Nov;23(13):1412-6. doi: 10.1177/0961203314540351. Epub 2014 Jun 24. PMID 24961747
- [Derived] Campos LM, Silva CA, Aikawa NE, Jesus AA, Moraes JC, Miraglia J, Ishida MA, Bueno C, Pereira RM, Bonfa E. High disease activity: an independent factor for reduced immunogenicity of the pandemic influenza a vaccine in patients with juvenile systemic lupus erythematosus. Arthritis Care Res (Hoboken). 2013 Jul;65(7):1121-7. doi: 10.1002/acr.21948. PMID 23818263
- [Derived] Miossi R, Fuller R, Moraes JC, Ribeiro AC, Saad CG, Aikawa NE, Miraglia JL, Ishida MA, Bonfa E, Caleiro MT. Immunogenicity of influenza H1N1 vaccination in mixed connective tissue disease: effect of disease and therapy. Clinics (Sao Paulo). 2013;68(2):129-34. doi: 10.6061/clinics/2013(02)oa02. PMID 23525305
- [Derived] Shinjo SK, de Moraes JC, Levy-Neto M, Aikawa NE, de Medeiros Ribeiro AC, Schahin Saad CG, Precioso A, Silva CA, Bonfa E. Pandemic unadjuvanted influenza A (H1N1) vaccine in dermatomyositis and polymyositis: immunogenicity independent of therapy and no harmful effect in disease. Vaccine. 2012 Dec 17;31(1):202-6. doi: 10.1016/j.vaccine.2012.10.063. Epub 2012 Oct 30. PMID 23123020
- [Derived] Aikawa NE, Campos LM, Goldenstein-Schainberg C, Saad CG, Ribeiro AC, Bueno C, Precioso AR, Timenetsky Mdo C, Silva CA, Bonfa E. Effective seroconversion and safety following the pandemic influenza vaccination (anti-H1N1) in patients with juvenile idiopathic arthritis. Scand J Rheumatol. 2013;42(1):34-40. doi: 10.3109/03009742.2012.709272. Epub 2012 Sep 20. PMID 22992045
- [Derived] Ribeiro AC, Laurindo IM, Guedes LK, Saad CG, Moraes JC, Silva CA, Bonfa E. Abatacept and reduced immune response to pandemic 2009 influenza A/H1N1 vaccination in patients with rheumatoid arthritis. Arthritis Care Res (Hoboken). 2013 Mar;65(3):476-80. doi: 10.1002/acr.21838. PMID 22949223
- [Derived] Guissa VR, Pereira RM, Sallum AM, Aikawa NE, Campos LM, Silva CA, Bonfa E. Influenza A H1N1/2009 vaccine in juvenile dermatomyositis: reduced immunogenicity in patients under immunosuppressive therapy. Clin Exp Rheumatol. 2012 Jul-Aug;30(4):583-8. Epub 2012 Aug 29. PMID 22931582
- [Derived] Franca IL, Ribeiro AC, Aikawa NE, Saad CG, Moraes JC, Goldstein-Schainberg C, Laurindo IM, Precioso AR, Ishida MA, Sartori AM, Silva CA, Bonfa E. TNF blockers show distinct patterns of immune response to the pandemic influenza A H1N1 vaccine in inflammatory arthritis patients. Rheumatology (Oxford). 2012 Nov;51(11):2091-8. doi: 10.1093/rheumatology/kes202. Epub 2012 Aug 20. PMID 22908326
- [Derived] Borba EF, Saad CG, Pasoto SG, Calich AL, Aikawa NE, Ribeiro AC, Moraes JC, Leon EP, Costa LP, Guedes LK, Silva CA, Goncalves CR, Fuller R, Oliveira SA, Ishida MA, Precioso AR, Bonfa E. Influenza A/H1N1 vaccination of patients with SLE: can antimalarial drugs restore diminished response under immunosuppressive therapy? Rheumatology (Oxford). 2012 Jun;51(6):1061-9. doi: 10.1093/rheumatology/ker427. Epub 2012 Jan 31. PMID 22298793
- [Derived] Aikawa NE, Campos LM, Silva CA, Carvalho JF, Saad CG, Trudes G, Duarte A, Miraglia JL, Timenetsky Mdo C, Viana VS, Franca IL, Bonfa E, Pereira RM. Glucocorticoid: major factor for reduced immunogenicity of 2009 influenza A (H1N1) vaccine in patients with juvenile autoimmune rheumatic disease. J Rheumatol. 2012 Jan;39(1):167-73. doi: 10.3899/jrheum.110721. Epub 2011 Nov 15. PMID 22089462
- [Derived] Ribeiro AC, Guedes LK, Moraes JC, Saad CG, Aikawa NE, Calich AL, Franca IL, Carvalho JF, Sampaio-Barros PD, Goncalves CR, Borba EF, Timenetsky Mdo C, Precioso AR, Duarte A, Bonfa E, Laurindo IM. Reduced seroprotection after pandemic H1N1 influenza adjuvant-free vaccination in patients with rheumatoid arthritis: implications for clinical practice. Ann Rheum Dis. 2011 Dec;70(12):2144-7. doi: 10.1136/ard.2011.152983. Epub 2011 Aug 22. PMID 21859696
- [Derived] Saad CG, Borba EF, Aikawa NE, Silva CA, Pereira RM, Calich AL, Moraes JC, Ribeiro AC, Viana VS, Pasoto SG, Carvalho JF, Franca IL, Guedes LK, Shinjo SK, Sampaio-Barros PD, Caleiro MT, Goncalves CR, Fuller R, Levy-Neto M, Timenetsky Mdo C, Precioso AR, Bonfa E. Immunogenicity and safety of the 2009 non-adjuvanted influenza A/H1N1 vaccine in a large cohort of autoimmune rheumatic diseases. Ann Rheum Dis. 2011 Jun;70(6):1068-73. doi: 10.1136/ard.2011.150250. PMID 21540203